CLINICAL TRIAL: NCT04767139
Title: Expanded Program for Immunization, a Missed Opportunity for Postpartum Family Planning Utilization: A Quasi Experimental Study
Brief Title: EPI, a Missed Opportunity for Postpartum Family Planning Utilization
Acronym: EPI
Status: Completed | Type: Observational
Sponsor: Hawassa University (Other)
Collaborators: EngenderHealth (Other)
Responsible Party: Principal Investigator, Abebaw Abeje Muluneh, Mr., Hawassa University
Other Study IDs: g6t4n7gi
Record Dates: First submitted 2021-02-19; First posted 2021-02-23 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Contraception
MeSH Terms: interventions — Counseling; Family Planning Services

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pre-intervention group: mothers included for the pre-intervention assessment of contraceptive prevalence rate in the selected health centers
- post intervention group: mothers included for the post-intervention assessment of contraceptive prevalence rate in the selected health centers
  Interventions: Behavioral: counseling for family planning

INTERVENTIONS:
Behavioral: counseling for family planning — all mothers presented to infant immunization units of the selected health centers will be counseled for family planning service and referred to the family planning unit if they decided to use.
  Groups: post intervention group

SUMMARY:
The global unmet need for postpartum family planning remains high, while immunization services are among the most widely utilized health services. Most women in the extended postpartum period want to delay or avoid future pregnancies but many are not using a modern contraceptive method. Establishing systematic screening, counseling, and referral systems from different contact points particularly from infant immunization units may improve family planning access and uptake in the extended postpartum period. Hence, this study is aimed to assess the effect of counseling for family planning at immunization units on postpartum contraceptive uptake during the extended postpartum period.

DETAILED DESCRIPTION:
Background: The global unmet need for postpartum family planning remains high, while immunization services are among the most widely utilized health services. Most women in the extended postpartum period want to delay or avoid future pregnancies but many are not using a modern contraceptive method. Establishing systematic screening, counseling, and referral systems from different contact points particularly from Expanded Program for Immunization (EPI) units may improve family planning access and uptake in the extended perinatal period.

Therefore, this study is proposed to assess the effect of counseling for family planning at immunization units on postpartum contraceptive uptake during the extended postpartum period.

To do this, a before-and-after type of quasi-experimental study will be conducted in purposively selected health centers in Sidama, South Ethiopia. All mothers coming to the selected health centers for infant immunization services will be screened for, counseled, and referred for family planning. A structured interviewer-administered questionnaire will be used to collect quantitative data from a total of 1474 randomly selected women coming to purposively selected health centers before and after the intervention. Bivariate and multivariable logistic regression analysis adjusting for possible confounding variables will be computed.

ELIGIBILITY:
Inclusion Criteria:

* all women visiting the selected health facilities at least two times during the pre-intervention period will be included

Exclusion Criteria:

* No exclussion critera

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Study Population: All women in the extended postpartum period visiting the selected health centers for infant immunization service are the study populations.
Sampling Method: Probability Sample
Enrollment: 1474 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-10-28 (Actual)

PRIMARY OUTCOMES:
improved contraceptive uptake | March 3, 2021
  the contraceptive utilization rate will be increased after the initiation of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Abebaw Abeje Muluneh, MSc, Principal Investigator — Hawassa University; Abel Gedefaw, MD, MPh, Study Chair — Hawassa University
Locations (1):
- Sidama regional health bureau, Awasa, Sidama Region, Ethiopia

REFERENCES:
- [Derived] Muluneh AA, Gedefaw A, Kelaye T, Sisay F, Worku M, Astatkie A, Shiferaw S. Addressing a missed opportunity for contraceptive use during the extended postpartum period by integrating it with infant immunization services in Sidama Region, Ethiopia: A quasi-experimental study. PLOS Glob Public Health. 2024 Jun 25;4(6):e0003236. doi: 10.1371/journal.pgph.0003236. eCollection 2024. PMID 38917099